CLINICAL TRIAL: NCT06834464
Title: Effect of Nanohydroxyapatite Paste After Different Pretreatment Techniques on Remineralization and Color Change of White Spot Lesions In Children: A Randomized Control Study.
Brief Title: Effect of Nanohydroxyapatite Paste After Different Pretreatment Techniques on White Spot White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Maryam Mohamed Ibrahim El Mansy, Researcher of Pediatric Dentistry, Orthodontics and Pediatric Dentistry Department, Oral and Dental Research Institute, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0343
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: White Spot Lesions
Keywords: white spot lesions; diagnodent; remineralization; nanohydroxyapatite
MeSH Terms: interventions — Hydrochloric Acid; Enamel Microabrasion

STUDY DESIGN:
Intervention Model Description: randomized controlled parallel double blinded study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding was done to the outcomes assessor and the child and care provider. the outcome assessor has assessed the outcome of each treatment without knowing the type of treatment done. the child was blinded as he was not aware of the type of treatment applied to him. The care provider was blind and he was not allowed to accompany the child during treatment application
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No treatment group (No Intervention): No treatment was applied (negative control)
- Nano hydroxyapatite paste group (Experimental): Nano hydroxyapatite paste was applied for 5 minutes
  Interventions: Drug: Nanohydroxyapatite paste
- HCl + Nano hydroxyapatite paste (Experimental): Pretreatment with 2% HCL for 20 sec then nano hydroxyapatite paste was applied for 5 minutes.
  Interventions: Drug: Nanohydroxyapatite paste; Drug: HCl liquid
- microabrasion + Nano hydroxyapatite paste (Experimental): Pretreatment with microabrasion with oplasture for 60 sec then nano hydroxyapatite paste was applied for 5 minutes.
  Interventions: Drug: Nanohydroxyapatite paste; Drug: microabrasion

INTERVENTIONS:
Drug: Nanohydroxyapatite paste — nanohydroxyapatite paste will be applied with a brush on the surface of the teeth
  Other Names: remineralizing paste
  Arms: HCl + Nano hydroxyapatite paste; Nano hydroxyapatite paste group; microabrasion + Nano hydroxyapatite paste
Drug: HCl liquid — HCl liquid will be applied for 60 seconds prior to application of nanohydroxyapatite paste in certain groups
  Other Names: hydrochloric acid
  Arms: HCl + Nano hydroxyapatite paste
Drug: microabrasion — the material will be applied on the surface of teeth then microabrasion will be done with a rubber cup for 60 seconds
  Other Names: opalasture
  Arms: microabrasion + Nano hydroxyapatite paste

SUMMARY:
forty teeth diagnosed with white spot lesions in children aged between 10-14 years old were selected to compare between the effect of using nanohydroxyapatite paste applicatio either alone or preceded by the application of HCl (hydrochloric acid) or microabrasion

DETAILED DESCRIPTION:
This study was designed as a randomized controlled double blinded clinical trial in which forty teeth clinically diagnosed with white spot lesions collected from children of both sexes with age range between 10-14 years old was selected from the outpatient clinics of the National Research Centre.

Ethical approval was obtained from the Medical Research Ethics Committee, National Research Centre with number 0343 Written informed consent was taken from the legal guardian of each participating child willing to participate in the trial, prior to the start of the clinical procedure after explaining the whole procedure in a simple way. The consent form was written in Arabic. verbal approval was taken from the child . Parallel allocation design was adopted for the intervention and control arms with allocation ration 1: 1 (i.e. 10 cases each).

The sample size was calculated considering the previously published studies with 80% power in detecting the true statistical significance among the four groups.

The inclusion criteria dictated that the patients should be in the age range of 10 to 14 years, presenting at least 1 White spot lesion on the labial surface of one or more permanent upper or lower anterior teeth.

The exclusion criteria involved patients who had hypoplastic enamel and those with dentine caries, patients who had systemic diseases and also uncooperative patients.

. All children involved in this study was instructed to brush their teeth under the supervision of the researcher before the application of the studied agent.

The buccal surfaces of the study-group teeth was cleaned with water slurry of pumice and rubber prophy cups. After cleaning and drying with a cotton roll, the application of the agent was done for 5 minutes using an applicator tip. After each application, children was instructed not to eat or drink for 1 hour

The same process was repeated in three separated visits in periods of one week, two weeks and six weeks on teeth in each of study and control group.

Grouping of samples:

Group 1: No treatment was applied (negative control). Group 2: Nano hydroxyapatite paste (Apagard primo toothpaste) was applied for 5 minutes.

Group 3: Pretreatment with 2% HCL for 20 sec then nano hydroxyapatite paste (Apagard primo toothpaste) was applied for 5 minutes.

Group 4: Pretreatment with microabrasion with oplasture for 60 sec then nano hydroxyapatite paste (Apagard primo toothpaste) was applied for 5 minutes.

Assessment:

A) Assessment of color change:

Color change of white spot lesions was assessed; before treatment, immediately after treatment, 2 weeks and 6 weeks after the onset of treatment on each tooth in each of study groups and control group using Vita easy shade device.

Prior each measurement, the device was calibrated according to the manufacturer's instructions.

B) Remineralization assessment:

Remineralization assessment was done using Laser fluorescence device "DIAGNOdent® (KaVo)".

All the teeth of the patients included in the study was examined using DIAGNOdent® (KaVo) as recommended by the manufacturer to assess the remineralization process.

All the measurements was performed using the Type B tip, which are designed for flat surfaces like the buccal one. Prior to each measurement, the device was calibrated using a ceramic standard according to the manufacturer's instructions.

The mineralization of the lesion was measured using DIAGNOdent laser fluorescence device before the application and another reading was recorded after 10 min of application. Other recordings was taken at one week, two weeks and six weeks on teeth in each of study and control group

ELIGIBILITY:
Inclusion criteria:

* age range of children is 10 to 14 years
* presence of at least 1 White spot lesion on the labial surface of one or more permanent upper or lower anterior teeth.

Exclusion criteria:

* hypoplastic enamel
* dentine caries,
* patients with systemic diseases
* uncooperative patient

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Assessment of color change | Color change of white spot lesions was assessed; before treatment, immediately after treatment, 2 weeks and 6 weeks after the onset of treatment on each tooth in each of study groups
  Color change of white spot lesions was assessed; the onset of treatment on each tooth in each of study groups and control group using Vita easy shade device.

SECONDARY OUTCOMES:
Remineralization assessment All the teeth of the patients included in the study will be examined using DIAGNOdent® (KaVo) as recommended by the manufacturer to assess the remineralization process. | Remineralization of white spot lesions was assessed; before treatment, immediately after treatment, 2 weeks and 6 weeks after the onset of treatment on each tooth in each of study groups
  Remineralization assessment was done using Laser fluorescence device "DIAGNOdent

CONTACTS AND LOCATIONS:
Overall Officials: Maryam m El Mansy, researcher, Principal Investigator — The National Research Centre, Egypt
Locations (1):
- the National research Centre, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to share

REFERENCES:
- [Background] Jayarajan J, Janardhanam P, Jayakumar P; Deepika. Efficacy of CPP-ACP and CPP-ACPF on enamel remineralization - an in vitro study using scanning electron microscope and DIAGNOdent. Indian J Dent Res. 2011 Jan-Feb;22(1):77-82. doi: 10.4103/0970-9290.80001. PMID 21525682
- [Background] Abou Neel EA, Aljabo A, Strange A, Ibrahim S, Coathup M, Young AM, Bozec L, Mudera V. Demineralization-remineralization dynamics in teeth and bone. Int J Nanomedicine. 2016 Sep 19;11:4743-4763. doi: 10.2147/IJN.S107624. eCollection 2016. PMID 27695330
- [Derived] El Mansy MM, Saleh RS, Rashed MF, El-Motayam AK. Effect of nanohydroxyapatite paste after different pretreatment techniques on remineralization and color change of white spot lesions in children: a randomized control study. BMC Oral Health. 2026 Jan 13. doi: 10.1186/s12903-025-07365-5. Online ahead of print. PMID 41530802